CLINICAL TRIAL: NCT02772614
Title: An Open-label Study in Healthy Male Subjects to Assess the Absorption, Distribution, Metabolism and Excretion of [14C]-Labelled BIA 3-202 and Metabolites Following a Single-dose Oral Administration
Brief Title: Absorption, Distribution, Metabolism and Excretion of [14C]-Labelled BIA 3-202 and Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-3202-106
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
Keywords: Nebicapone, Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — nebicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nebicapone (200 mg) (Experimental): Each subject was to receive one single dose of 2.5 MBq [14C]-labelled BIA 3-202 (200 mg) together with a total of 250 mL non-carbonated water.
  The study drug was given after an overnight fast of at least 10 hours after the in-house stay. During waking hours on Day 1, subjects had to have a fluid intake of at least 150 mL per hour starting 1 hour before study drug administration.
  Interventions: Drug: BIA 3-202 (200 mg)

INTERVENTIONS:
Drug: BIA 3-202 (200 mg) — 200 mg powder for oral use of unlabelled BIA 3-202

SUMMARY:
The purpose of this study is:

To determine the rate and routes of excretion of BIA 3-202 and the mass balance in urine and faeces To determine the kinetics of total radioactivity in blood To determine the kinetics of total radioactivity in plasma To determine the kinetics of BIA 3-202 and its metabolites in plasma

DETAILED DESCRIPTION:
Monocentre, open, non-placebo-controlled, single-group, single-dose study. Safety measurements (12-lead ECG, vital signs, blood chemistry and haematology) were conducted before and after the study, adverse events were monitored throughout the study.

Each subject was to receive a single oral dose of 2.5 MBq [14C]-labelled BIA 3-202 (200 mg). This was the intended radiolabelled dose without any losses; the actual administered dose was of 2.29 MBq [14C]-labelled BIA 3-202 (200 mg). Subjects were hospitalized the day before the administration until 264 hours thereafter.

Whole blood samples (2 mL) for total radioactivity analysis, plasma samples (1.5 mL) for total radioactivity analysis, and plasma samples (7 mL) for analysis of BIA 3-202 and its metabolites were collected at the following times: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, and 264 hours post-dose.

Urine was sampled before the drug administration (pre-dose), then it was collected from 0-4, 4-8, 8-24, 24-48, 48-72, 72-120, 120-168, 168-216, and 216-264 hours post-dose.

Aliquots of each sample were taken for liquid scintillation counting by the investigator.

Aliquots were separated for determination of parent drug and metabolite patterns.

A baseline faeces sample was obtained during the screening or baseline period. Following dose, each faeces sample was collected in a separate container during the 264 hours post-dose period.

Vomitus (if produced) was collected.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, 40-55 years of age. Take only Caucasians.
2. Clinically acceptable sitting blood pressure and pulse rate , i.e.: BP: 110-160 mmHg systolic, 65-95 mmHg diastolic and pulse rate: 50-100 bpm. Blood pressure and pulse will be measured after 3 minutes resting in a sitting position.
3. Subject body weight must be between 50 and 95 kg and within -10% / +20% of normal for their height and frame size (according to Metropolitan Life Insurance Table, see Appendix 1&2 of the Study Protocol). Frame size will be determined using elbow breadth measurement.
4. Normal 12-lead ECG.
5. Ability to communicate well with the investigator and comply with the requirements of the entire study.
6. The subject has given his written informed consent to participate in the study.

Exclusion Criteria:

1. History of serious adverse reactions or hypersensitivity to any drug.
2. Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
3. History of alcohol or drug abuse in the last 5 years.
4. Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
5. Need of any prescription medication within 14 days prior to the administration of the drug and/or nonprescription medication within 7 days prior to the administration of the drug.
6. Participation in other clinical trials during the previous month in which an investigational drug or a commercially available drug was tested.
7. Loss of 500 mL blood or more during the 3 month period before the study, e.g., as a donor.
8. Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e., impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhoea or conditions associated with total or partial obstruction of the urinary tract.
9. Symptoms of a significant somatic or mental illness in the 4 week period preceding drug administration.
10. History of hepatitis B and / or C and / or positive serology results which indicate the presence of hepatitis B and / or C.
11. Positive results from the HIV serology.
12. Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation, however, liver parameters (SGPT, SGOT) and CK values must be within the normal range.
13. Positive results of the drug screening.
14. Known hypersensitivity to BIA 3-202.
15. Heavy smokers, i.e., more than 10 cigarettes per day.
16. Exposure to artificial ionizing radiation in the last 12 months (e.g., x-ray investigation).
17. Subject who had more than 4 flights (with more than 2 hours flight time) within the last year prior to the administration of the drug.

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2006-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration (Cmax) | pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, and 264 hours post-dose
time of occurrence of Cmax (tmax) | pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, and 264 hours post-dose
area under the plasma concentration-time curve from time zero to the last sampling time at which concentrations are at or above the limit of quantification, calculated by the linear trapezoidal rule (AUC0-t) | pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, and 264 hours post-dose
area under the plasma concentration versus time curve from time zero to infinity, calculated from AUC0-t + (C(t)/λz), where C(t) is the last quantifiable concentration and λz the apparent terminal rate constant (AUC0-∞) | pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, and 264 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Pharma Contract Ltd, Allschwil, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No